CLINICAL TRIAL: NCT00997763
Title: Randomized Comparison of Everolimus- Eluting Stent Versus Sirolimus-Eluting Stent Implantation for De Novo Coronary Artery DisEase in Patients With DIABETES Mellitus
Brief Title: Comparison of Everolimus-Eluting Stent vs Sirolimus-Eluting Stent in Patients With DIABETES Mellitus
Acronym: ESSENCE-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0220
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
Keywords: stenting, XIENCE V, CYPHER
MeSH Terms: conditions — Coronary Artery Disease; Cardiomyopathy, Dilated, 1C

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XIENCE V (Active Comparator): everolimus-eluting stent
  Interventions: Device: XIENCE V
- CYPHER (Active Comparator): Using Cypher stent
  Interventions: Device: CYPHER

INTERVENTIONS:
Device: XIENCE V — everolimus-eluting stent
  Other Names: Xience V stent
  Arms: XIENCE V
Device: CYPHER — sirolimus-eluting stent
  Other Names: Cypher elect stent
  Arms: CYPHER

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of coronary stenting with the Everolimus- Eluting stent compared to the Sirolimus-Eluting stent in the treatment of de novo coronary stenosis in patients with diabetic patients.

DETAILED DESCRIPTION:
Diabetic patients often present unfavorable coronary anatomy with small and diffusely diseased vessels (1) and exhibit exaggerated neointimal hyperplasia after bare-metal stent (BMS) implantation as compared with nondiabetics (2). Although drug-eluting stent (DES) implantation significantly reduced the neointimal hyperplasia and angiographic restenosis compared to BMS in diabetic patients (3), presence of diabetes mellitus (DM) have been still associated with an increased risk of restenosis and unfavorable clinical outcomes in the era of DES (4,5). Recently, the relative efficacies of sirolimua-eluting stent (SES) and paclitaxel-eluting stent (PES) in patients with DM have been evaluated in randomized and registry studies (6-10). The present study, ESSENCE-DIABETES Study, compare 8-month angiographic and 1-year clinical outcomes in patients with diabetes mellitus treated with sirolimus-eluting stent (CYPHER) or everolimus-eluting stent (XIENCE V)

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with angina and documented ischemia or patients with documented silent ischemia
* Patients who are eligible for intracoronary stenting
* Age >18 years, <75 ages
* De novo lesion
* Percent diameter stenosis ≥50%
* Reference vessel size ≥ 2.5 mm by visual estimation

Exclusion Criteria:

* History of bleeding diathesis or coagulopathy
* Pregnant state
* Known hypersensitivity or contra-indication to contrast agent and heparin
* Limited life-expectancy (less than 1 year)
* Acute ST elevation myocardial infarction on admission
* Characteristics of lesion

  1. Left main disease
  2. In-stent restenosis
  3. Graft vessels
* Hematological disease (Neutropenia <3000/mm3, Thrombocytopenia <100,000/mm3)
* Hepatic dysfunction, liver enzyme (ALT and AST) elevation ≥ 3 times normal
* Renal dysfunction, creatinine ≥ 2.0mg/dL
* Contraindication to aspirin, clopidogrel or cilostazol
* Left ventricular ejection fraction <30%
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Angiographic in-segment late loss at angiography | 8-month

SECONDARY OUTCOMES:
All-cause Death | 12 month
All-cause Death | 5 year
Cardiac death | 12 months
Cardiac death | 5 year
Myocardial infarction | 12 months
Myocardial infarction | 5 year
Target vessel revascularization (all and ischemia-driven) | 12 months
Target lesion revascularization (all and ischemia-driven) | 5 year
Stent thrombosis by definition of Academic Research Consortium (ARC) | 12 months
Stent thrombosis by definition of Academic Research Consortium (ARC) | 5 year
Binary restenosis in both in-stent and in-segment | 8 months
Angiographic pattern of restenosis | 8 months

CONTACTS AND LOCATIONS:
Locations (18):
- South Korea (18):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Busan Saint Mary's Hospital, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Cheongju Saint Mary's Hospital, Cheongju-si
  - Kangwon University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Daejeon St Mary's Hospital Catholic University, Daejeon
  - Asan Medical Center, Gangneung
  - Chonbuk National University Hospital, Jeonju
  - Kyungsang University Hospital, Jinju
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan Natioanal University Hospital, Pusan
  - Hallym University Sacred Heart Hospital, Pyeongchon
  - Asan Medical Center, Seoul
  - Hallym University Sacred Heart Hospital, Seoul
  - Korea Veterans Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.